CLINICAL TRIAL: NCT02286895
Title: An Evaluation of the Immune Response to Pentavalent Rotavirus Vaccine After a Supplemental Dose Given at 9 Months of Age With Local EPI Vaccines in Mali
Brief Title: Immune Response to Rotavirus Vaccine After a Supplemental Dose Given at 9 Months of Age With Local EPI Vaccines in Mali
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: PATH (Other)
Collaborators: Center for Vaccine Development - Mali (Other); University of Maryland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PATH-RVI-PRV-01
Record Dates: First submitted 2014-10-01; First posted 2014-11-10 (Estimated); Results first posted 2018-12-07 (Actual); Last update posted 2019-01-02 (Actual); Status verified 2018-12

CONDITIONS: Diarrhea Rotavirus
Keywords: rotavirus; rotavirus vaccine; Mali; EPI vaccines
MeSH Terms: interventions — RotaTeq; Measles Vaccine; Yellow Fever Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (without rotavirus vaccine) (Active Comparator): Group A will receive measles vaccine (MV), yellow fever vaccine (YFV), and meningitis conjugate vaccine (PsA-TT-5μg).
  Interventions: Biological: measles vaccine (MV); Biological: yellow fever vaccine (YFV); Biological: meningitis conjugate vaccine (PsA-TT-5μg)
- Group B (with rotavirus vaccine) (Experimental): Group A will receive measles vaccine (MV), yellow fever vaccine (YFV), and meningitis conjugate vaccine (PsA-TT-5μg) plus one oral dose of pentavalent rotavirus vaccine (PRV).
  Interventions: Biological: pentavalent rotavirus vaccine (PRV); Biological: measles vaccine (MV); Biological: yellow fever vaccine (YFV); Biological: meningitis conjugate vaccine (PsA-TT-5μg)

INTERVENTIONS:
Biological: pentavalent rotavirus vaccine (PRV) — Each two-ml dose contains 5 live human-bovine reassortant rotaviruses with a minimum of 2.0 - 2.8 x 106 infectious units (IU) per reassortant, depending on the serotype, and not greater than 116 x 106 IU per aggregate dose. Each vaccine dose contains sucrose, sodium citrate, sodium phosphate monobasic monohydrate, sodium hydroxide, polysorbate 80, cell culture media, and trace amounts of fetal bovine serum. RotaTeq contains no preservatives. RotaTeq is a pale yellow clear liquid that may have a pink tint. This vaccine was administered orally.
  Other Names: RotaTeq
  Arms: Group B (with rotavirus vaccine)
Biological: measles vaccine (MV) — A lyophilized vaccine in a pack containing one vial plus one ampoule of sterile water for injection. After reconstitution, each 0.5 ml/dose of MV contains active substances not less than 1000 units of 50% cell culture infectious doses (CCID50) of MV. Measles Vaccine Live Attenuated virus is propagated on Human Diploid Cells. This MV is currently part of the local EPI program in Mali. This vaccine was administered subcutaneously to the right deltoid.
Biological: yellow fever vaccine (YFV) — A freeze-dried live attenuated yellow fever virus of the 17D strain for injection. After reconstitution, one dose (0.5 ml) contains active substances not less than 1000 units of 50% lethal doses (LD50) of yellow fever virus. This YFV is currently part of the local EPI program in Mali. This vaccine was administered intramuscularly to the left deltoid.
Biological: meningitis conjugate vaccine (PsA-TT-5μg) — A meningococcal A vaccine, with meningococcal A polysaccharide (PsA) conjugated to the carrier protein, tetanus toxoid (TT). After reconstitution, one dose (0.5 ml) contains 5μg meningococcal A polysaccharide and 5-16 μg tetanus toxoid as a carrier protein. PsA-TT-5μg was considered experimental at the initiation of this study, but received approval from the WHO for infants on 30 December 2014. For all participants enrolled January 1st, 2015 or later, PsA-TT-5μg was not included in Group A or Group B, due to its December 2014 expiration date. This vaccine was administered intramuscularly to the right thigh.
  Other Names: PsA-TT

SUMMARY:
This study is an evaluation of the immune response to pentavalent rotavirus vaccine (PRV) after an additional fourth dose is given at 9 months of age with local World Health Organization (WHO) Expanded Programme on Immunization (EPI) vaccines in Mali.

DETAILED DESCRIPTION:
Vaccination is the best way to prevent severe rotavirus disease and the deadly, dehydrating diarrhea that it causes. However, given only moderate efficacy in the first year of life and a possible further decline in immunity, it is considered a top priority by public health experts to evaluate the possible value of a "booster" dose of rotavirus vaccine in low income countries to confer longer duration of protection into the second year of life when disease burden continues to be high.

This study is an open-label, individual-randomized, parallel-group, comparative immunogenicity trial. Participating infants randomized to Group A will receive one dose each of measles vaccine (MV), yellow fever vaccine (YFV), and meningitis conjugate vaccine (PsA-TT-5μg) at 9 months of age, and infants randomized to Group B will receive one dose each of MV, YFV, PsA-TT-5μg, and PRV at 9 months of age.

The study will simultaneously evaluate two primary objectives, one for noninferiority of the response to MV given with PRV (co-primary objective 1) and one for noninferiority of the response to YFV given with PRV (co-primary objective 2).

Secondary objectives of the study were the following:

1. To evaluate the non-inferiority of the immune response 3 months post-vaccination (as sero-conversion) to MV given with PRV (Group B) to that given without PRV (Group A).
2. To compare the immune response (as geometric mean titers [GMTs]) to YFV given with PRV (Group B) to that given without PRV (Group A).
3. To evaluate the non-inferiority of the immune response (as sero-response) to PsA-TT-5μg given with PRV (Group B) compared to that given without PRV (Group A).
4. To compare the immune response (as GMTs) to PsA-TT-5μg given with PRV (Group B) to that given without PRV (Group A).
5. To evaluate the superiority of the immune response (as sero-response and geometric mean concentrations [GMCs]) to a supplemental dose of PRV given at 9 months of age with local EPI vaccines (Group B) compared no supplemental dose (Group A).
6. To describe the safety profile of study vaccination with PRV.

ELIGIBILITY:
Inclusion Criteria:

* At least 9 months of age through 11 months of age (has not yet reached 1st birthday) at the time of administration of study vaccines.
* Residence in the study area.
* At least one parent or guardian who is at least 18 years of age and is willing to provide written informed consent.
* Generally healthy and free of obvious health problems as established by medical history including physical examination and clinical judgment of the investigator.
* A child who is fully vaccinated according to the local EPI schedule (exclusive of oral polio vaccine birth dose).
* A parent or guardian is willing to attend all planned study visits or allow home visits and mobile phone contacts, as required by the protocol.

Exclusion Criteria:

* Previous receipt any measles-containing vaccine.
* Previous receipt of any yellow fever vaccine.
* Previous receipt of any meningitis vaccine.
* Receipt of rotavirus vaccine within the past 90 days.
* Administration of any other vaccine within 8 weeks prior to administration of study vaccines or planned vaccination during the 4 weeks after study vaccination.
* History of allergic disease or known hypersensitivity to any component of the study vaccines and/or following administration of vaccines included in the local program of immunization
* Use of any investigational or non-registered drug within 90 days prior to the administration of study vaccines.
* Administration of immunoglobulins and/or any blood products within 90 days prior to the administration of study vaccines or planned administration during the vaccine period.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying agents since birth (including systemic corticosteroids, this means prednisone, or equivalent, ≥0.5 mg/kg/day; topical steroids including inhaled steroids are allowed).
* A family history of congenital or hereditary immunodeficiency.
* History of intussusception.
* Uncorrected congenital malformation of the gastrointestinal tract that would predispose for intussusception.
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic, or renal functional abnormality, as determined by medical history or physical examination, which in the opinion of the investigator, might interfere with the study objectives.
* Acute illness at the time of enrollment (acute disease is defined as the presence of a moderate or severe illness with fever [axillary temperature ≥38°C] or without fever [severity determined at the discretion of the investigator]. Acute illness is a temporary exclusion.
* Any condition or criterion that in the opinion of the investigator might compromise the well-being of the subject or the compliance with study procedures or interfere with the outcome of the study.

Ages: 9 Months to 11 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 600 (Actual)
Dates: Start 2014-10; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samba O Sow, MD, Msc, Principal Investigator — Center for Vaccine Development - Mali
Locations (1):
- CVD-Mali, Bamako, Mali

REFERENCES:
- [Derived] Haidara FC, Tapia MD, Sow SO, Doumbia M, Coulibaly F, Diallo F, Traore A, Kodio M, Kelly CL, Fitzpatrick M, Kotloff K, Victor JC, Neuzil K. Evaluation of a Booster Dose of Pentavalent Rotavirus Vaccine Coadministered With Measles, Yellow Fever, and Meningitis A Vaccines in 9-Month-Old Malian Infants. J Infect Dis. 2018 Jul 13;218(4):606-613. doi: 10.1093/infdis/jiy215. PMID 29659924

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited up to 750 healthy male and female infant subjects of 9-11 months of age from the local communities and community health centers in Bamako, Mali. The duration of planned study participation for each subject was to be approximately 3 months and the estimated duration of the recruitment period was to be 3 months.
Groups:
- Group A (Without Rotavirus Vaccine): Group A will receive measles vaccine (MV), yellow fever vaccine (YFV), and meningitis conjugate vaccine (PsA-TT-5μg).
  measles vaccine (MV): At enrollment, all infants will receive one dose of 0.5ml subcutaneously
  yellow fever vaccine (YFV): At enrollment, all infants will receive one dose of 0.5ml intramuscularly
  meningitis conjugate vaccine (PsA-TT-5μg): At enrollment, all infants will receive one dose of 0.5ml intramuscularly
- Group B (With Rotavirus Vaccine): Group A will receive measles vaccine (MV), yellow fever vaccine (YFV), and meningitis conjugate vaccine (PsA-TT-5μg) plus one oral dose of pentavalent rotavirus vaccine (PRV).
  pentavalent rotavirus vaccine (PRV): At enrollment, infants in this group receive one dose of 2.0ml orally
  measles vaccine (MV): At enrollment, all infants will receive one dose of 0.5ml subcutaneously
  yellow fever vaccine (YFV): At enrollment, all infants will receive one dose of 0.5ml intramuscularly
  meningitis conjugate vaccine (PsA-TT-5μg): At enrollment, all infants will receive one dose of 0.5ml intramuscularly
Period: Randomized and Vaccinated
Arm/Group | Group A (Without Rotavirus Vaccine) | Group B (With Rotavirus Vaccine)
Started | 300 | 300
Completed | 300 | 300
Not Completed | 0 | 0
Period: Assessed for Measles Seroconversion
Arm/Group | Group A (Without Rotavirus Vaccine) | Group B (With Rotavirus Vaccine)
Started | 300 | 300
Completed | 252 | 261
Not Completed | 48 | 39
Not completed — Protocol Violation | 1 | 4
Not completed — Missing measurement | 6 | 3
Not completed — Baseline measure non-negative | 41 | 32

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A (Without Rotavirus Vaccine) | Group B (With Rotavirus Vaccine) | Total
Number analyzed (Participants) | 300 | 300 | 600
Age, Continuous [Mean (Standard Deviation); unit: months] | 9.7 (.7) | 9.7 (.7) | 9.7 (.7)
Age, Customized [Count of Participants; unit: Participants]
  9 months | 223 | 224 | 447
  10 months | 53 | 51 | 104
  11 months | 24 | 25 | 49
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 133 | 151 | 284
  Male | 167 | 149 | 316
Region of Enrollment [Number; unit: participants]
  Mali | 300 | 300 | 600
Ethnicity [Count of Participants; unit: Participants]
  Bambara | 101 | 120 | 221
  Mandika/Malinke | 41 | 37 | 78
  Fula/Peulh | 49 | 34 | 83
  Sarahule/Sarakole | 35 | 37 | 72
  Other | 74 | 72 | 146

OUTCOME MEASURES:

1. Primary Outcome: Number/Percentage of Subjects With Seroconversion for Anti-measles Immunoglobulin G (IgG) Antibody
Description: Measured using a commercially-available Enzyme Linked Immunosorbent Assay (ELISA). Seroconversion was defined as a measurement ≥1.10 geometric mean titer (GMT) at Day 28 among subjects with measurement ≤0.90 at baseline
Time Frame: 28 days post-vaccination
Population: Number of subjects with valid measurements and measurement ≤0.90 at baseline (per protocol)
Measure: Count of Participants; unit: Participants
Arm/Group | Group A (Without Rotavirus Vaccine) | Group B (With Rotavirus Vaccine)
Number analyzed (Participants) | 252 | 261
Participants
  Seroconversion | 246 | 255
  No seroconversion (≤0.90) | 2 | 3
  Equivocal measurements (≥0.91 and ≤1.09) | 4 | 3
Statistical Analysis 1: Comparison: Group A (Without Rotavirus Vaccine) vs Group B (With Rotavirus Vaccine); Based on results from a prior study, the sponsor assumed 90% sero-conversion rates in each Arms A and B for each antigen in the two co-primary objectives. To rule out a non-inferiority margin of no more than 10% with 95% power (95% power was chosen to give an overall power of at least 90%) and a one-sided type-one error rate of no more than 2.5%, 237 evaluable subjects were required in each group to explore the co-primary objectives; Test type: Non-Inferiority — The protocol stated that non-inferiority would be achieved if the lower limit of the 95% confidence interval (2-sided) for the difference in sero-conversion percentages (group receiving rotavirus minus group not receiving rotavirus) was > -10%; Mean Difference (Net) = 0.1, 95% CI 2-sided [-4.0 to 4.2]

2. Primary Outcome: Number/Percentage of Subjects With Seroresponses for Yellow Fever Neutralizing Antibody
Description: Measured by virus neutralization assay, determined using Robert Koch Institute's yellow fever standard of practice and relative to international scientific references for which the level of anti-YF neutralizing IgG protection was known. Seroresponse was defined as a geometric mean titer (GMT) of at least four times baseline value.
Time Frame: 28 days post-vaccination
Population: Number of subjects with valid measurements and negative result at baseline (per protocol)
Measure: Count of Participants; unit: Participants
Arm/Group | Group A (Without Rotavirus Vaccine) | Group B (With Rotavirus Vaccine)
Number analyzed (Participants) | 290 | 287
Participants
  Seroresponse | 153 | 141
  No seroresponse | 137 | 146
Statistical Analysis 1: Comparison: Group A (Without Rotavirus Vaccine) vs Group B (With Rotavirus Vaccine); Based on results from a prior study completed by PATH and CVD-Mali, the sponsor assumed 90% sero-conversion rates in each Arms A and B for each antigen in the two co-primary objectives. To rule out a non-inferiority margin of no more than 10% with 95% power (95% power was chosen to give an overall power of at least 90%) and a one-sided type-one error rate of no more than 2.5%, 237 evaluable subjects were required in each group to explore the co-primary objectives; Test type: Non-Inferiority — The protocol stated that non-inferiority would be achieved if the lower limit of the 95% CI (2-sided) for the difference in sero-conversion percentages (group receiving rotavirus minus group not receiving rotavirus) was > -10%; Mean Difference (Net) = -4.1, 95% CI 2-sided [-12.2 to 4.0]

3. Secondary Outcome: Number/Percentage of Subjects With Seroconversion for Anti-measles Immunoglobulin G (IgG) Antibody
Description: as for outcome 1
Time Frame: 3 months post-vaccination
Population: Subjects with valid measurements and measurement ≤0.90 at baseline (per protocol)
Measure: Count of Participants; unit: Participants
Arm/Group | Group A (Without Rotavirus Vaccine) | Group B (With Rotavirus Vaccine)
Number analyzed (Participants) | 218 | 228
Participants
  Seroconversion | 206 | 210
  No seroconversion (≤0.90) | 4 | 5
  Equivocal measurements (≥0.91 and ≤1.09) | 8 | 13
Statistical Analysis 1: Comparison: Group A (Without Rotavirus Vaccine) vs Group B (With Rotavirus Vaccine); [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Mean Difference (Net) = -2.4, 95% CI 2-sided [-7.5 to 2.7]

4. Secondary Outcome: Serum Neutralization Geometric Mean Titers for Yellow Fever Vaccine
Description: Measured by virus neutralization assay, determined using Robert Koch Institute's yellow fever standard of practice (SOP) and relative to international scientific references for which the level of anti-YF neutralizing IgG protection was known.
Time Frame: 28 days post-vaccination
Population: Number of subjects with valid measurements (per protocol)
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group A (Without Rotavirus Vaccine) | Group B (With Rotavirus Vaccine)
Number analyzed (Participants) | 293 | 293
titer
  Baseline | 2.4 [2.3 to 2.5] | 2.5 [2.4 to 2.6]
  28 days post-vaccination | 16.8 [14.8 to 19.1] | 15 [13.3 to 17.0]
Statistical Analysis 1: Comparison: Group A (Without Rotavirus Vaccine) vs Group B (With Rotavirus Vaccine); Test type: Equivalence — Definition of equivalence/null hypothesis: geometric mean titer (GMT) of group receiving rotavirus vaccine divided by GMT of group not receiving rotavirus vaccine = 1; geometric mean titer ratio = 0.9, 95% CI 2-sided [0.8 to 1.1]

5. Secondary Outcome: Number/Percentage of Subjects With Seroresponses for Meningitis Conjugate Serum Bactericidal Antibody (SBA)
Description: Seroresponse was defined as a geometric mean titer (GMT) of at least four times baseline value. Measured using baby rabbit complement (rSBA).
Time Frame: 28 days post-vaccination
Population: Number of subjects with valid measurements (per protocol)
Measure: Count of Participants; unit: Participants
Arm/Group | Group A (Without Rotavirus Vaccine) | Group B (With Rotavirus Vaccine)
Number analyzed (Participants) | 293 | 292
Participants
  Seroresponse | 276 | 273
  No seroresponse | 17 | 19
Statistical Analysis 1: Comparison: Group A (Without Rotavirus Vaccine) vs Group B (With Rotavirus Vaccine); Test type: Equivalence — Definition of equivalence/null hypothesis: geometric mean concentration (GMC) of group receiving rotavirus vaccine/ GMC of group not receiving rotavirus vaccine = 1; geometric mean titer ratio = -0.7, 95% CI 2-sided [-5.2 to 3.8]

6. Secondary Outcome: Geometric Mean of Meningitis Serum Bactericidal Antibody Titer
Description: Measured using baby rabbit complement (rSBA).
Time Frame: Baseline to Day 28
Population: Number of subjects with valid measurements (per protocol)
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group A (Without Rotavirus Vaccine) | Group B (With Rotavirus Vaccine)
Number analyzed (Participants) | 293 | 292
titer | 2.8 [2.4 to 3.3] | 3.2 [2.7 to 3.9]
Statistical Analysis 1: Comparison: Group A (Without Rotavirus Vaccine) vs Group B (With Rotavirus Vaccine); Test type: Equivalence — [test comment as in outcome 4, analysis 1]; geometric mean titer ratio = 0.9, 95% CI 2-sided [0.7 to 1.3]

7. Secondary Outcome: Number/Percentage of Subjects With Anti-rotavirus Immunoglobulin A (IgA) Titer at Least 3 Times Baseline Value
Description: Conducted by validated Enzyme Linked Immunosorbent Assay (ELISA). The pre- and post-vaccination samples were to be evaluated in one run for consistency and each specimen was to be tested with a negative control for better specificity.
Time Frame: 28 days post-vaccination
Population: Number of subjects with valid measurements (per protocol)
Measure: Count of Participants; unit: Participants
Arm/Group | Group A (Without Rotavirus Vaccine) | Group B (With Rotavirus Vaccine)
Number analyzed (Participants) | 292 | 292
Participants
  At least 3 times baseline value | 80 | 131
  Not at least 3 times baseline value | 212 | 161
Statistical Analysis 1: Comparison: Group A (Without Rotavirus Vaccine) vs Group B (With Rotavirus Vaccine); Null hypothesis: percentage of the seroresponse to rotavirus in the group that received rotavirus vaccine minus the percentage of the seroresponse to rotavirus in the group that did not receive rotavirus vaccine is less than or equal to 0; Test type: Superiority; Mean Difference (Net) = 17.5, 95% CI 2-sided [9.7 to 25.3]

8. Secondary Outcome: Number/Percentage of Subjects With Anti-rotavirus IgA Titer of ≥20 Units/mL
Description: as for outcome 7
Time Frame: 28 days post-vaccination
Population: Number of subjects with valid measurements (per protocol)
Measure: Count of Participants; unit: Participants
Arm/Group | Group A (Without Rotavirus Vaccine) | Group B (With Rotavirus Vaccine)
Number analyzed (Participants) | 292 | 292
Participants
  ≥20 Units/mL | 172 | 218
  <20 Units/mL | 120 | 74
Statistical Analysis 1: Comparison: Group A (Without Rotavirus Vaccine) vs Group B (With Rotavirus Vaccine); [analysis description as in outcome 7, analysis 1]; Test type: Superiority; Mean Difference (Net) = 15.8, 95% CI 2-sided [8.1 to 23.4]

9. Secondary Outcome: Number/Percentage of Subjects With Anti-rotavirus IgA <20 Units/mL at Baseline Visit That Had >=20 Units/mL at Day 28
Description: as for outcome 7
Time Frame: 28 days post-vaccination
Population: Participants with valid measures of anti-rotavirus IgA <20 units/mL at baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Group A (Without Rotavirus Vaccine) | Group B (With Rotavirus Vaccine)
Number analyzed (Participants) | 165 | 160
Participants
  Seroresponse | 52 | 91
  No seroresponse | 113 | 69
Statistical Analysis 1: Comparison: Group A (Without Rotavirus Vaccine) vs Group B (With Rotavirus Vaccine); [analysis description as in outcome 7, analysis 1]; Test type: Superiority; Mean Difference (Net) = 25.4, 95% CI 2-sided [14.6 to 36.2]

10. Secondary Outcome: Number/Percentage of Subjects With Anti-rotavirus IgG Titer at Least 3 Times Baseline Value
Description: as for outcome 7
Time Frame: 28 days post-vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | Group A (Without Rotavirus Vaccine) | Group B (With Rotavirus Vaccine)
Number analyzed (Participants) | 293 | 293
Participants
  Seroresponse | 77 | 168
  No seroresponse | 216 | 125
Statistical Analysis 1: Comparison: Group A (Without Rotavirus Vaccine) vs Group B (With Rotavirus Vaccine); [analysis description as in outcome 7, analysis 1]; Test type: Superiority; Mean Difference (Net) = 31.1, 95% CI 2-sided [23.1 to 39.0]

11. Secondary Outcome: Number/Percentage of Subjects With Anti-rotavirus IgG Titer of ≥20 Units/mL
Description: as for outcome 7
Time Frame: 28 days post-vaccination
Population: Number of subjects with valid measurements (per protocol)
Measure: Count of Participants; unit: Participants
Arm/Group | Group A (Without Rotavirus Vaccine) | Group B (With Rotavirus Vaccine)
Number analyzed (Participants) | 293 | 293
Participants
  ≥20 Units/mL | 223 | 275
  <20 Units/mL | 70 | 18
Statistical Analysis 1: Comparison: Group A (Without Rotavirus Vaccine) vs Group B (With Rotavirus Vaccine); [analysis description as in outcome 7, analysis 1]; Test type: Superiority; Mean Difference (Net) = 17.7, 95% CI 2-sided [12.0 to 23.5]

12. Secondary Outcome: Number/Percentage of Subjects With Anti-rotavirus IgG <20 Units/mL at Baseline Visit That Had >=20 Units/mL at Day 28
Description: as for outcome 7
Time Frame: 28 days post-vaccination
Population: Participants with valid measures of anti-rotavirus IgA <20 units/mL at baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Group A (Without Rotavirus Vaccine) | Group B (With Rotavirus Vaccine)
Number analyzed (Participants) | 92 | 91
Participants
  Seroresponse | 29 | 76
  No seroresponse | 63 | 15
Statistical Analysis 1: Comparison: Group A (Without Rotavirus Vaccine) vs Group B (With Rotavirus Vaccine); [analysis description as in outcome 7, analysis 1]; Test type: Superiority; Mean Difference (Net) = 52.0, 95% CI 2-sided [37.7 to 66.3]

13. Secondary Outcome: Geometric Mean of Anti-rotavirus IgA Concentration
Description: as for outcome 7
Time Frame: 28 days post-vaccination
Population: Number of subjects with valid measurements (per protocol)
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group A (Without Rotavirus Vaccine) | Group B (With Rotavirus Vaccine)
Number analyzed (Participants) | 292 | 292
titer
  Baseline | 23.7 [18.6 to 30.3] | 25.3 [19.7 to 32.6]
  28 days post-vaccination | 67.9 [49.9 to 92.3] | 118.4 [90.9 to 154.3]
Statistical Analysis 1: Comparison: Group A (Without Rotavirus Vaccine) vs Group B (With Rotavirus Vaccine); Null hypothesis: geometric mean titer (GMT) in group receiving rotavirus vaccine/GMT in group not receiving rotavirus vaccine ≤ 1; Test type: Superiority; geometric mean titer ratio = 1.7, 95% CI 2-sided [1.2 to 2.4]

14. Secondary Outcome: Geometric Mean of Anti-rotavirus IgG Concentration
Description: as for outcome 7
Time Frame: 28 days post-vaccination
Population: Number of subjects with valid measurements (per protocol)
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group A (Without Rotavirus Vaccine) | Group B (With Rotavirus Vaccine)
Number analyzed (Participants) | 293 | 293
titer
  Baseline | 58.9 [47.1 to 73.7] | 62.5 [49.6 to 78.8]
  28 days post-vaccination | 153.3 [113.8 to 206.5] | 363.6 [293.6 to 450.4]
Statistical Analysis 1: Comparison: Group A (Without Rotavirus Vaccine) vs Group B (With Rotavirus Vaccine); Null hypothesis: 28 days post-vaccination, geometric mean titer (GMT) in group receiving rotavirus vaccine/GMT in group not receiving rotavirus vaccine ≤ 1; Test type: Superiority; geometric mean titer ratio = 2.3, 95% CI 2-sided [1.7 to 3.1]

15. Secondary Outcome: Geometric Mean of Anti-rotavirus IgA Among Subjects With <20 Units/mL Concentration at Baseline
Description: as for outcome 7
Time Frame: 28 days post-vaccination
Measure: Mean (95% Confidence Interval); unit: titer
Arm/Group | Group A (Without Rotavirus Vaccine) | Group B (With Rotavirus Vaccine)
Number analyzed (Participants) | 165 | 160
titer
  Baseline | 5.1 [4.7 to 5.5] | 4.8 [4.4 to 5.1]
  28 days post-vaccination | 22.2 [15.2 to 32.6] | 41.5 [29.8 to 57.9]
Statistical Analysis 1: Comparison: Group A (Without Rotavirus Vaccine) vs Group B (With Rotavirus Vaccine); [analysis description as in outcome 13, analysis 1]; Test type: Superiority; geometric mean titer ratio = 2.0, 95% CI 2-sided [1.2 to 3.3]

16. Secondary Outcome: Geometric Mean of Anti-rotavirus IgG Among Subjects With <20 Units/mL Concentration at Baseline
Description: as for outcome 7
Time Frame: 28 days post-vaccination
Population: Participants with valid measures of anti-rotavirus IgG <20 units/mL at baseline
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group A (Without Rotavirus Vaccine) | Group B (With Rotavirus Vaccine)
Number analyzed (Participants) | 92 | 91
titer
  Baseline | 7.8 [6.9 to 8.9] | 7.4 [6.5 to 8.4]
  28 days post-vaccination | 28.3 [16.3 to 49.2] | 123.7 [83.1 to 184.2]
Statistical Analysis 1: Comparison: Group A (Without Rotavirus Vaccine) vs Group B (With Rotavirus Vaccine); [analysis description as in outcome 13, analysis 1]; Test type: Superiority; geometric mean titer ratio = 4.6, 95% CI 2-sided [2.4 to 8.9]

17. Secondary Outcome: Number/Percentage of Participants Experiencing Immediate Reactions Post-vaccination
Description: With emphasis on allergic reactions, observed by study staff
Time Frame: Within 30 minutes post-vaccination
Population: Among all subjects enrolled (intent-to-treat population)
Measure: Count of Participants; unit: Participants
Arm/Group | Group A (Without Rotavirus Vaccine) | Group B (With Rotavirus Vaccine)
Number analyzed (Participants) | 300 | 300
Participants
  Any immediate reaction | 0 | 0
  No immediate reaction | 300 | 300

18. Secondary Outcome: Number of Solicited Adverse Reactions (AR) Experienced by Participants
Description: identified or observed by study staff during home visits and/or reported by a parent at any time. Solicited adverse reactions were graded and sub-categorized as those deemed related to vaccination or not by the investigator.
Time Frame: 7 days post-vaccination
Measure: Count of Units; unit: systemic reaction
Units Other Than Participants: systemic reaction
Arm/Group | Group A (Without Rotavirus Vaccine) | Group B (With Rotavirus Vaccine)
Number analyzed (Participants) | 300 | 300
Number analyzed (systemic reaction) | 41 | 38
systemic reaction
  Diarrhea | 24 | 21
  Vomiting | 8 | 7
  Pyrexia | 5 | 8
  Irritability | 1 | 2
  Lethargy | 2 | 0
  Rash | 1 | 0

19. Secondary Outcome: Number/Percentage of Participants Experiencing Serious Adverse Events (SAE)
Description: Occurring from vaccination through 3 months post-vaccination, identified or observed by study staff and/or reported by a parent at any time. Serious adverse events were graded for severity and sub-categorized as those deemed related to vaccination or not by the investigator.
Time Frame: 3 months post-vaccination
Population: Among all subjects enrolled (intent-to-treat population)
Measure: Count of Participants; unit: Participants
Arm/Group | Group A (Without Rotavirus Vaccine) | Group B (With Rotavirus Vaccine)
Number analyzed (Participants) | 300 | 300
Participants
  At least 1 SAE probably related to vaccination | 1 | 0
  At least 1 SAE not related to vaccination | 6 | 7
  No SAE | 292 | 293
  1 SAE unlikely to be related to vaccination | 1 | 0

ADVERSE EVENTS:
Time Frame: 3 months post-vaccination (death and serious adverse events), 28 days (all other adverse events)
Description: Field staff members visited study subjects on Days 1 through 5 to inquire about specific local and systemic signs and symptoms. On Day 7, a physician visited the subject's home for evaluation. Subjects returned to the study center on Day 28 and Day 84 for evaluation. After Day 28, only SAEs (with the exception of signs of potential intussusception) did not require documentation. A malaria test was conducted on Days 0, 28, and 84.
Arm/Group | Group A (Without Rotavirus Vaccine) | Group B (With Rotavirus Vaccine)
All-Cause Mortality (participants affected / at risk) | 0/300 | 0/300
Serious Adverse Events (participants affected / at risk) | 8/300 | 7/300
Other Adverse Events (participants affected / at risk) | 125/300 | 103/300
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A (Without Rotavirus Vaccine) (N=300) | Group B (With Rotavirus Vaccine) (N=300)
Gastroenteritis (Gastrointestinal disorders) | 2 | 2
Bronchitis (Infections and infestations) | 2 | 0
Malaria (Infections and infestations) | 1 | 5
Pharyngitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Burns second degree (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (Without Rotavirus Vaccine) (N=300) | Group B (With Rotavirus Vaccine) (N=300)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Otitis media (Ear and labyrinth disorders) | 1 | 0
Otitis media acute (Ear and labyrinth disorders) | 5 | 6
Otorrhoea (Ear and labyrinth disorders) | 1 | 0
Conjunctivitis (Eye disorders) | 3 | 2
Diarrhoea (Gastrointestinal disorders) | 41 | 30
Gastroenteritis (Gastrointestinal disorders) | 12 | 6
Vomiting (Gastrointestinal disorders) | 8 | 7
Irritability (General disorders) | 1 | 2
Lethargy (General disorders) | 2 | 0
Pyrexia (General disorders) | 5 | 8
Allergic respiratory symptoms (Immune system disorders) | 32 | 21
Bronchitis (Infections and infestations) | 1 | 3
Candida infection (Infections and infestations) | 1 | 0
Conjunctivitis bacterial (Infections and infestations) | 1 | 0
Ear infection (Infections and infestations) | 0 | 1
Impetigo (Infections and infestations) | 3 | 0
Malaria (Infections and infestations) | 7 | 7
Nasopharyngitis (Infections and infestations) | 6 | 8
Pharyngitis (Infections and infestations) | 4 | 5
Rhinitis (Infections and infestations) | 61 | 55
Staphylococcal skin infection (Infections and infestations) | 2 | 2
Varicella (Infections and infestations) | 1 | 0
Impetigo (Infections and infestations) | 2 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1
Wound (Injury, poisoning and procedural complications) | 1 | 1
Bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No